CLINICAL TRIAL: NCT07129135
Title: The Effect of Methylene Blue Bladder Instillation Versus No Intervention on Urinary Tract Injuries During Cesarean Hysterectomy for Placenta Accreta Spectrum: A Randomized Controlled Trial
Brief Title: Effect of Methylene Blue Bladder Instillation on Urinary Tract Injuries During Cesarean Hysterectomy for Placenta Accreta Spectrum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Usama Ahmed Elsaeed Salem, MD (Other)
Responsible Party: Sponsor-Investigator, Usama Ahmed Elsaeed Salem, MD, MD, Lecturer of Obstetrics and Gynecology, Faculty of Medicine, Cairo University., Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MD-316-2021
Record Dates: First submitted 2025-08-04; First posted 2025-08-19 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Placenta Accreta Spectrum; Abnormal Placentation; Cesarean Hysterectomy; Urinary Tract Injury; Bladder Injury
Keywords: Placenta Accreta Spectrum; Cesarean Hysterectomy; Methylene Blue; Bladder Filling; Bladder Injury; Ureteric Injury; Surgical Complications
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group, Methylene Blue Group, (Filled bladder Group) (Experimental)
  Interventions: Procedure: The bladder was filled with 300 ml diluted methylene blue (in normal saline) via Foley's catheter
- Control Group, Standard Care Group, (Not filled bladder Group) (No Intervention)

INTERVENTIONS:
Procedure: The bladder was filled with 300 ml diluted methylene blue (in normal saline) via Foley's catheter — The bladder was filled with 300 ml diluted methylene blue (in normal saline) via Foley's catheter before uterine incision or bladder dissection to help determine the borders better and enable dissection of the lower uterine segment without excessive bleeding or unintended Bladder kept distended during dissection.
  Arms: Intervention Group, Methylene Blue Group, (Filled bladder Group)

SUMMARY:
This randomized controlled trial aims to evaluate whether preoperative bladder filling with methylene blue dye can reduce the incidence of urinary tract injuries during cesarean hysterectomy in patients diagnosed with placenta accreta spectrum. A total of 60 patients will be randomly assigned to either an intervention group receiving methylene blue bladder instillation or a control group receiving standard surgical care. The primary outcome is the rate of intraoperative urinary tract injuries. Secondary outcomes include total operative time, , and pre and post operative hemoglobin level , number of units of packed RBCs transfused, number of units of fresh frozen plasma transfused, number of participants admitted to ICU postoperatively,number of participants with postoperative complications, duration of hospital stay of participants.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years
* Pregnant women diagnosed antenatally with placenta accreta spectrum (PAS).
* Pregnant women with history of previous one or more caesarian deliveries .
* Planned cesarean hysterectomy at ≥33 weeks of gestation.
* Singleton pregnancy.
* BMI <35 kg/m²
* Suitable for standardized General anaesthesia

Exclusion Criteria:

* Previous bladder surgery or known urologic abnormalities.
* Bleeding tendency disorder
* Renal failure .
* Allergy to methylene blue dye.
* Emergency hysterectomy without time for protocol preparation.
* Conservative uterine- preservation management.
* Refusal or inability to provide informed written consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-22 (Actual); Primary Completion 2025-01-05 (Actual); Study Completion 2025-01-25 (Actual)

PRIMARY OUTCOMES:
Number and percentage of patients with intraoperative urinary tract injuries (bladder, ureters). | Intraoperative (Day 0) to 24 hours post operatively.
  Number and percentage of patients with bladder or ureteric injury confirmed intraoperatively by direct visualization or intraoperative dye testing.

SECONDARY OUTCOMES:
Preoperative Hemoglobin recorded in g/dl | within 24 hours before surgery
  Venous sample obtained within 24 hours before surgery;Analyzed using the hospital's hematology analyzer; results recorded in g/dL.
Total number of Units of Packed Red Blood Cells (PRBC) Transfused | from surgery start to 24 hours postoperatively
  Total units from surgery start to 24 hours postoperatively, following a standardized transfusion protocol based on predefined hemoglobin thresholds, hemodynamic status, and coagulation parameters.
Total number of Units of Fresh Frozen Plasma (FFP) Transfused | from surgery start to 24 hours postoperatively
  Total units from surgery start to 24 hours postoperatively, given for abnormal coagulation (PT/aPTT >1.5× normal), suspected coagulopathy, or massive transfusion activation.
Total Operative time (minutes) | Measured in minutes from skin incision to closure.
Postoperative Hemoglobin recorded in g/dl | within 24 hours after surgery completion
  Venous sample obtained within 24 hours after surgery completion; earlier if major bleeding or hemodynamic instability occurred. Same analyzer used for consistency.
Number and percentage of patients admitted to ICU postoperatively. | Postoperatively during hospital stay up to 14 days postoperative.
Number of participants with postoperative complications | From time of surgery until hospital discharge (up to 14 days).
  Postoperative complications were recorded for each participant from the time of surgery until hospital discharge. Complications included pelvic hematoma and whether or not need relaparotomy , urinoma , thromboembolic events, ileus, and any other clinically significant adverse events documented in the patient's chart
Post operative hospital stay : Number of days from surgery to discharge . | Number of days from surgery to discharge (up to 14 days).
  Number of days of hospital stay from surgery to discharge (up to 14 days).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months after publication of study results for a year.
Access Criteria: Data will be shared upon reasonable request by contacting the corresponding author. Researchers must sign a data use agreement to access the data.